CLINICAL TRIAL: NCT05314920
Title: Cost-effectiveness of Transdiagnostic Group Psychological Treatment for Common Mental Disorders in Primary Care (PsicAP-Costs2): a Randomized Controlled Clinical Trial
Brief Title: Cost-effectiveness of a Transdiagnostic Psychological Treatment for Emotional Disorders in Primary Care
Acronym: PsicAP-Costs2
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Instituto de Investigación Marqués de Valdecilla (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: PsicAP-Costs2
Record Dates: First submitted 2022-01-25; First posted 2022-04-07 (Actual); Last update posted 2022-05-20 (Actual); Status verified 2022-05

CONDITIONS: Emotional Disorder
Keywords: transdiagnostic therapy; emotional disorders; primary care; cost-benefit analysis; brief psychological treatments; cognitive behavioral therapy; randomized controlled trial; depression; anxiety disorders; somatoform disorders
MeSH Terms: conditions — Depression; Anxiety Disorders; Somatoform Disorders

STUDY DESIGN:
Intervention Model Description: Multicenter randomized controlled trial with pre-post measures and 12-month follow-up.
Who Masked: Participant
Masking Description: Outcomes assessors will be blinded during pre- and post-treatment. Participants will be blinded during pretreatment assessment; however, it cannot be guaranteed that they will keep blinded in post-treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- transdiagnostic cognitive-behavioural therapy (TD-CBT) (Experimental): Transdiagnostic cognitive-behavioral group therapy: The psychological interventions will be manualized. Patients assigned to the experimental group will receive 7 sessions (1.5 hr/session) in groups of approximately 8-10 individuals over a 12-week period.
  Interventions: Behavioral: Transdiagnostic cognitive-behavioral therapy (TD-CBT)
- relaxation therapy (Active Comparator): The control group will receive a progressive muscle relaxation group intervention, based on the Bernstein and Borkoveck procedure. Patients will receive 7 sessions (1.5 hr/session) in groups of 8-10 individuals over a 12-week period.
  Interventions: Behavioral: Bernstein and Borkovec progressive muscle relaxation (PMR)

INTERVENTIONS:
Behavioral: Transdiagnostic cognitive-behavioral therapy (TD-CBT) — Transdiagnostic cognitive-behavioral therapy (TD-CBT)
  Arms: transdiagnostic cognitive-behavioural therapy (TD-CBT)
Behavioral: Bernstein and Borkovec progressive muscle relaxation (PMR) — Bernstein and Borkovec progressive muscle relaxation (PMR)
  Arms: relaxation therapy

SUMMARY:
The aim of this study is to test the cost-effectiveness and cost-utility of adding a transdiagnostic group cognitive-behavioural therapy (TD-CBT) to treatment as usual (TAU) for emotional disorders in primary care . A single-blind randomized controlled clinical trial will be conducted to compare the TD-CBT group therapy plus TAU to progressive muscle relaxation (PMR) group plus TAU in individuals, aged 18 to 65, with emotional disorders in four primary care centres located in Cantabria, Spain. The study will take a societal perspective. Psychological assessments will be carried out at baseline, post-treatment, and 12-months follow-up. The assessments will include measures of clinical symptoms (anxiety, depression, and/or somatic), dysfunction, cognitive-emotional factors (ruminative processes, pathological concern, attentional and interpretative biases, emotion regulation strategies and meta-cognitive beliefs), and satisfaction with the treatment received. Data on health service use, including medication and days of absence from work, will be collected from electronic medical records. The primary outcomes are the incremental cost-effectiveness ratios (ICER) based on the difference in mean costs and effectiveness between interventions and incremental cost-utility ratios (ICURs) based on health-related quality of life at post-treatment and 12-month follow-up. Secondary outcome measures include clinical symptoms, quality of life, functioning and treatment satisfaction. Bootstrap sampling will be used to assess the uncertainty of the results. Secondary moderation and mediation analyses will also be conducted. In addition, in sessions' number 1, 4 and 7 of both treatment arms, two questionnaires will be administered that collect therapeutic alliance and group satisfaction. The main study hypothesis is that adding TD-CBT to TAU in primary care will be more cost-effective than TAU plus PMR. In addition, these gains will be maintained in the 12-month follow-up. If it is successful, the dissemination of cost-effective treatment can help to overcome problems in accessing psychological treatment for emotional disorders in the context of an increasing demand for mental healthcare in primary care.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 to 65, inclusive, who present to the PC centre seeking treatment for anxiety, depressive or somatic symptoms.
* Scores above the predetermined cut-off points on the GAD-7 (>= 10), the PHQ-9 (>= 10) or the PHQ-15 (>=10 plus a score of 2 in three or more somatic symptoms).
* Agreement to participate in the study, with written informed consent.

Exclusion Criteria:

* Major depressive disorder (PHQ-9> 24) and/or severe disability (SDS > 25) will be interviewed by a clinician for the presence of any severe mental disorder, including autism spectrum disorders, bipolar disorder, schizophrenia, anorexia nervosa, substance dependence, personality disorder.
* Presence of severe or recent suicide attempts
* Presence of intellectual disability (IQ < 70).
* Be receiving psychological treatment or any type of specialized care related to mental health.
* Insufficient Spanish language skills

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
Change in cost-effectiveness data | Baseline, immediately after the intervention, and 12-month follow-up
  Cost-effectiveness results will be calculated by the ICER, defined as the difference in mean costs between interventions divided by the difference in their effectiveness according to the symptom questionnaires' mean scores.
  The healthcare data collected will be used for cost calculations. To calculate healthcare-related costs, an ad hoc questionnaire will be used to collect emotional disorder-related healthcare data (public and private healthcare consultations, accidents, medical tests, and sick leaves in the past 3 months; psychotropic drugs or other medication, and their posology).
Change in cost-utility data | Baseline, immediately after the intervention, and 12 month follow-up
  Cost-utility will be measured through the healthcare data collected above and the European Quality of Life Scale (EuroQoL, EQ) (The EuroQol Group, 1990), calculating the QALYS and the ICURs, defined as the difference in mean cost divided by the difference in mean QALYs. The Spanish version of the 5-domain, 5-level EuroQol (EQ-5D-5L) (Badia et al., 1999; van Reenen et al., 2019) will be used to assess health status in five dimensions (mobility, self-care, daily activities, pain/unease, and anxiety/depression) with five levels of severity (no problems, slight problems, moderate problems, severe problems, and either extreme problems or unable to perform activity).

SECONDARY OUTCOMES:
Change in depressive symptoms: Patient Health Questionnaire - 9 item (PHQ-9) | Baseline, immediately after the intervention, and 12 month follow-up
  The PHQ-9 (Kroenke et al., 2001) is the depression module of the PHQ (Díez-Quevedo et al., 2001; Spitzer et al., 1999) that scores the 9 DSM-IV depression criteria in the last two weeks. Is a nine item, self-report scale that ranges from 0 to 27 (higher scores means a worse outcome).
Change in anxiety symptoms: Generalized Anxiety Disorder - 7 item (GAD-7) | Baseline, immediately after the intervention, and 12 month follow-up
  The GAD-7 (Spitzer et al., 2006) assesses common anxiety symptoms in the last two weeks. It is composed of seven self-report items ranging from 0 to 21 points. Higher scores means a greater presence of anxiety symptoms.
Change in somatic symptoms: Patient Health Questionnaire - 15 item (PHQ-15) | Baseline, immediately after the intervention, and 12 month follow-up
  The PHQ-15 (Kroenke et al., 2002) is the somatization module of the PHQ and scores symptoms present in the past four weeks. The scale is composed of fifteen self-report items, ranging from 0 to 30. Higher scores means a worse outcome.
Change in functioning: Sheehan Disability Scale (SDS) | Baseline, immediately after the intervention, and 12 month follow-up
  The SDS (Sheehan et al., 1996) is a five item self-reported scale composed of three main domains (work, family and social functioning) and two optional items (perceived stress and perceived social support). It ranges from 0 to 50, with higher scores indicating a worse outcome.
Change in treatment satisfaction | Immediately after the intervention and 12-month follow-up
  Posttreatment and 12-month follow-up assessments will also collect an additional question about treatment satisfaction, through a Likert-type question, ranging from 0 to 10.

OTHER OUTCOMES:
Change in rumination: Ruminative Responses Scales (brooding subscale) (RRS-B) | Baseline, immediately after the intervention, and 12-month follow-up
  The RRS-B (Nolen-Hoeksema & Morrow, 1991) is composed of five self-reported items, ranging from 5 to 20. Higher scores means a worse outcome.
Change in worry: Penn State Worry Questionnaire - Abbreviated (PSWQ-A) | Baseline, immediately after the intervention, and 12-month follow-up
  The PSWQ-A (Meyer et al., 1990) measures the pathological worry as an uncontrollable and general state. The scale is composed of eight self-reported items, ranging from 5 to 40. Higher scores means a worse outcome
Change in attentional and interpretative biases: Inventory of Cognitive Activity in Anxiety Disorders (IACTA) | Baseline, immediately after the intervention, and 12-month follow-up
  The IACTA was originally developed by Cano-Vindel (2001). It includes subscales that assess distortions according to Eysenck's four-factor theory (Eysenck, 2000). The scale is composed of five self-reported items, ranging from 0 to 20. Higher scores means a worse outcome.
Change in emotion regulation: Cognitive Emotion Regulation Questionnaire (CERQ) | Baseline, immediately after the intervention, and 12-month follow-up
  The CERQ-36 (Garnefski et al., 2001) was developed for measuring the specific cognitive emotion regulation strategies that a person uses to face a stressful event (self-blame, acceptance, rumination, positive refocus, refocus on planning, positive reappraisal, putting into perspective, catastrophizing or blaming others). It scores from 1 ("almost never") to 5 ("almost always") how often the participant thinks as described. The 27-item shortened version will be used (Holgado-Tello et al., 2018). Each cognitive strategy is assessed by means of three items, ranging from 3 to 15. Higher scores means a greater use of the strategy.
Change in metacognitive beliefs: Metacognitions Questionnaire (negative beliefs subscale) (MCQ) | Baseline, immediately after the intervention, and 12-month follow-up
  The MCQ-NB (Wells & Cartwright-Hatton, 2004) is a short form of the original MCQ (Cartwright-Hatton & Wells, 1997), which measures the beliefs about the own thinking processes. The scale is composed of six self-reported items, ranging from 6 to 24. Higher scores means a worse outcome.
Change in cognitive Distortions in Emotional Disorders (CDTE) | Baseline, immediately after the intervention, and 12-month follow-up
  The CDTE (The PsicAP Group, unpublished) measures the frequency of certain cognitive biases. It includes sixteen self-reported items that measure the presence of four factors: sustained attention bias, divided attention bias, magnification interpretational bias, and catastrophization interpretational bias. It ranges from 0 to 4. Higher scores means a greater presence of the cognitive bias.
Change in alliance: Working Alliance Inventory Patient Form (WAI-P) and Group Session Rating Scale (GSRS) | In therapy sessions number 1, 4 and 7
  The WAI-P (Andrade-González & Fernández-Liria, 2015) is a thirty-six self-report scale that measure perceived therapeutic alliance. It ranges from 36 to 252 with higher scores indicating better alliance between patient and clinical professional.
  The GSRS (Duncan & Miller, 2007) is a four self-reported scale that assess alliance to the group. It ranges from 0 to 40, with higher scores indicating better alliance between the patient and the group of therapy.

CONTACTS AND LOCATIONS:
Locations (4):
- Spain (4):
  - Centro Sanitario "Sardinero", Santander
  - Centro Sanitario "Dávila", Santander
  - Centro Sanitario "Camargo Costa", Santander
  - Centro Sanitario "Camargo Interior", Santander

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gonzalez-Blanch C, Barrio-Martinez S, Priede A, Martinez-Gomez S, Perez-Garcia-Abad S, Miras-Aguilar M, Ruiz-Gutierrez J, Munoz-Navarro R, Ruiz-Rodriguez P, Medrano LA, Prieto-Vila M, Carpallo-Gonzalez M, Aguilera-Martin A, Galvez-Lara M, Cuadrado F, Moreno E, Garcia-Torres F, Vencesla JF, Corpas J, Jurado-Gonzalez FJ, Moriana JA, Cano-Vindel A. Cost-effectiveness of transdiagnostic group cognitive behavioural therapy versus group relaxation therapy for emotional disorders in primary care (PsicAP-Costs2): Protocol for a multicentre randomised controlled trial. PLoS One. 2023 Mar 16;18(3):e0283104. doi: 10.1371/journal.pone.0283104. eCollection 2023. PMID 36928238